CLINICAL TRIAL: NCT05635214
Title: Real Time Remote Tele-Mentored Ultrasonography to Assist Emergency Medicine Providers at Physician Shortage Designation Hospitals
Brief Title: Real Time Remote Tele-Mentored Ultrasonography in the ED
Acronym: ED RTMUS
Status: Withdrawn | Type: Observational
Why Stopped: Poor community engagement
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Alexis Salerno, Assistant Professor of Emergency Medicine, University of Maryland, Baltimore
Other Study IDs: HP-00104001
Record Dates: First submitted 2022-11-08; First posted 2022-12-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Abdominal Pain; Flank Pain
Keywords: ultrasound; telemedicine; emergency medicine
MeSH Terms: conditions — Abdominal Pain; Flank Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with RUQ or Flank Pain: These are patients who present to the emergency department with abdominal pain or flank pain.
  Interventions: Procedure: real time remote tele mentored ultrasound exam

INTERVENTIONS:
Procedure: real time remote tele mentored ultrasound exam — A patient will have a point of care ultrasound exam performed by a local provider with a remote expert guiding them through the exam using video conferencing.

SUMMARY:
The goal of this pilot study is to evaluate the use of real time remote tele-mentored ultrasound in the emergency department at hospitals with physician shortage designation. The main question the investigators aim to answer is:

• Will RTMUS be used in instances where it is available and indicated for abdominal pain or flank pain.

DETAILED DESCRIPTION:
Point-of-care-ultrasound (POCUS) decreases time for clinical diagnosis and improves provider diagnostic accuracy. The use of the Focused Assessment with Sonography in Trauma (FAST) has decreased time to surgical intervention by over 50% for hypotensive trauma patients. POCUS also improves resource utilization, reducing the 6-month ionizing radiation exposure in patients with suspected renal colic in one study. Despite advances in deploying POCUS, the remaining gap is an adequate number of emergency department providers who feel confident in performing POCUS examinations, limiting the delivery of healthcare services to patients at the point of care. Real time remote tele-mentored ultrasound (RTMUS) can overcome this practice gap by enabling remote ultrasound experts to provide real-time assistance to bedside providers using a telemedicine platform. Preliminary studies at the investigator's institution have demonstrated the feasibility of deploying RTMUS to guide nurses in the intensive care setting to acquire accurate images suitable for complex clinical decision making. In this preliminary study, RTMUS had good concordance (90%-100%) between radiological transthoracic echocardiography or CT for evaluating cardiac findings such as left ventricular function, right ventricular dysfunction and pericardial effusion. The overall objective of this study is to examine the impact of RTMUS integration to emergency departments in hospitals with physician shortage designations. The investigators hypothesize the RTMUS system will be able to provide images sufficient for clinical diagnosis and that the local ED providers will accept RTMUS as a suitable option for ultrasound.

User's Acceptability of RTMUS: In this aim, the investigators will evaluate emergency department user's acceptability of RTMUS for abdominal pain and flank pain. The investigators hypothesize that in eligible patients, RTMUS will be used in at least 10% of the instances in which it is available and indicated. As a secondary data point, stakeholder surveys will be collected on the use and performance of RTMUS.

RTMUS is an innovative solution that can improve patient care. This project will engage emergency department providers at physician shortage designation hospitals to increase the use of POCUS in their clinical practice. In the future, RTMUS can be applied to various resource constrained settings to help providers use POCUS to care for their patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the emergency department with abdominal pain or flank pain.
* Age greater than or equal to 18 years

Exclusion Criteria:

* Patients who do not present to the emergency department with abdominal pain or flank pain.
* Age less than 18 years
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: -Patients who present to the emergency department with abdominal pain or flank pain.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with abdominal pain or flank pain in which RTMUS is used | through study completion, an average of 6 months
  ED patients with chief complaint of abdominal pain or flank pain

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Salerno, MD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: No